CLINICAL TRIAL: NCT06757894
Title: Efficacy and Safety of Zuberitamab and Bendamustine Combination Treatment Followed by Monotherapy Maintenance in Treatment-naïve Follicular Lymphoma: an Open-label, Prospective, Multicenter, Single-arm Phase II Clinical Study
Brief Title: Efficacy and Safety of Zuberitamab Combined with Bendamustine, Followed by Monotherapy Maintenance, in Treatment-naïve Follicular Lymphoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Gansu Cancer Hospital (Other); Ganzhou Cancer Hospital (Unknown); Fifth Affiliated Hospital, Sun Yat-Sen University (Other); Fifth Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2024-815-01
Record Dates: First submitted 2024-12-27; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Follicular Lymphoma (FL)
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Zuberitamab and Bendamustine Combination Treatment (Experimental): Induction therapy:
  1. Zuberitamab: 375 mg/m², administered on Day 1 (D1) of Cycles 1-6 (C1-C6).
  2. Bendamustine: 90 mg/m², administered on D1-2 of C1-C6. Each cycle lasts 28 days. After 6 cycles of treatment, patients who achieve complete remission (CR) or partial remission (PR) will continue with maintenance therapy.
  Maintenance therapy:
  Zuberitamab: 375 mg/m², administered once every 2 months, until disease progression or for a maximum of 24 months (12 doses).
  Interventions: Drug: Zuberitamab; Drug: Bendamustine

INTERVENTIONS:
Drug: Zuberitamab — 375 mg/m², administered on Day 1 (D1) of Cycles 1-6 (C1-C6)
Drug: Bendamustine — 90 mg/m², administered on D1-2 of C1-C6

SUMMARY:
This is a prospective, single-arm, multicenter, phase ll clinical trial to evaluate the efficacy and safety of Zuberitamab and Bendamustine combination treatment in treatment-naïve follicular lymphoma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signing of informed consent.
2. Age ≥ 18 years, no gender restriction.
3. Histologically confirmed follicular lymphoma (grades 1-3a), CD20 positive by immunohistochemistry.
4. No prior systemic treatment for FL.
5. Ann Arbor stage III/IV, or stage II with bulky disease (bulky disease defined as a tumor diameter ≥ 7 cm).
6. Presence of measurable lesions.
7. Meeting any of the following criteria:

   1. B symptoms: unexplained fever >38°C, night sweats, unexplained weight loss >10% in the last 6 months.
   2. Abnormal signs: splenomegaly, pleural effusion, ascites, etc.
   3. Major organ damage: involvement of major organs leading to organ dysfunction.
   4. Hematologic involvement: cytopenia [WBC < 1.0 × 10⁹/L and/or PLT < 100 × 10⁹/L]; leukemia-like manifestations (malignant cells > 5.0 × 10⁹/L); elevated LDH levels; HGB < 120 g/L; β2-microglobulin ≥ 3 mg/L.
   5. Bulky disease: involvement of ≥ 3 tumors with each diameter ≥ 3 cm, or any lymph node or extranodal tumor with diameter ≥ 7 cm (for Ann Arbor stage III-IV patients).
   6. Tumor enlargement of 20%-30% within 2-3 months, or approximately 50% enlargement within 6 months.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
9. Expected survival of > 6 months.

Exclusion Criteria:

1. History of allergy to any component of monoclonal antibodies or investigational drugs.
2. Central nervous system involvement.
3. History of previous malignant tumors.
4. Clinically significant cardiac or pulmonary diseases.
5. Infection requiring intravenous antibiotic treatment or hospitalization within 4 weeks prior to enrollment; or infection requiring oral antibiotics within 2 weeks prior to enrollment; or symptoms related to an infection within 1 week prior to enrollment.
6. Major surgery within 4 weeks prior to enrollment.
7. Vaccination with live vaccines within 4 weeks prior to enrollment or planned live vaccination during the study.
8. HIV antibody positive.
9. Active syphilis infection, TP antibody positive, and anti-TP treatment within the last 2 years.
10. Hepatitis C virus (HCV) antibody positive with HCV RNA quantitative test result exceeding the detection limit; Hepatitis B surface antigen (HBsAg) positive or Hepatitis B core antibody (HBcAb) positive, with Hepatitis B virus DNA quantitative test result exceeding the detection limit (for patients with HBsAg or HBcAb positive status, regardless of HBV-DNA detection, oral entecavir or other antiviral therapy must be initiated prior to enrollment and continued according to the physician's instructions during the trial).
11. Pregnant or breastfeeding women, or planning to become pregnant during the study.
12. Investigator determines the patient is unsuitable for enrollment or may not be able to complete the trial for other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2034-02-01 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) | Up to 6 cycles (each cycle is 28 days).
  Defined as the proportion of patients who achieve complete remission at the end of induction therapy.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 6 cycles (each cycle is 28 days).
  The proportion of patients who achieve complete remission (CR) or partial remission (PR) at the end of induction therapy.
Progression-Free Survival (PFS) | From the start of induction therapy to the first documented disease progression or death from any cause, whichever occurs first, assessed up to 78 months.
  The length of time during and after treatment that a patient lives with cancer without it getting worse or progressing.
Event-Free Survival (EFS) | From the start of induction therapy to the first occurrence of any event, including disease progression, discontinuation of treatment, or death for any reason, whichever occurs first, assessed up to 78 months.
  The length of time during and after treatment during which a patient remains free from any of the following events: disease progression, treatment discontinuation for any reason, or death from any cause.
Duration of Response (DOR) | From the first documentation of CR or PR to the first documented disease progression, assessed up to 78 months.
  The length of time during and after treatment that a patient's disease remains under control or in remission. It is the period from the first documentation of a response (such as partial or complete remission) until disease progression or relapse occurs.
Overall Survival (OS) | From the start of induction therapy to death from any cause, assessed up to 78 months.
  The length of time from the date of enrollment until death from any cause.
Time to Next Treatment (TTNT) | From the start of induction therapy to the start of the next line of anti-tumor treatment, assessed up to 78 months.
  The length of time from the initiation of a current treatment until the patient requires a subsequent line of therapy for the cancer.
Incidence and severity of Adverse Events (AE) and Serious Adverse Event (SAE) | From the start of induction therapy through the end of the maintenance therapy phase, up to 30 months.
  The occurrence and intensity of undesirable or harmful effects experienced by patients associated with the use of a medical treatment or intervention during the clinical trial.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Universitiy Cancer Center, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided